CLINICAL TRIAL: NCT00164125
Title: An Open Label Study of Chronic Polyethyleneglycol3350 Use in Constipated Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 851-CR3
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

INTERVENTIONS:
Drug: polyethyleneglycol3350

SUMMARY:
To evaluate the safety of extended use of polyethyleneglycol3350 laxative in constipated patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Male or female outpatients at least 18 years of age
* Constipated according to ROME I criteria
* If female and of childbearing potential, patient must be surgically sterilized or using oral contraceptives, depot contraceptives, intrauterine device, or testifies that she is monogamous with a vasectomized partner, or practices abstinence and will continue to do so during the duration of study
* Are otherwise in good health, as judged by a physical examination
* In the investigator's judgment, patient is mentally competent to sign an instrument of informed consent

Exclusion Criteria:

* Patients with heme positive stool at screening. Patients with heme positive stool that can be attributed to hemorrhoids or anal fissures are eligible for inclusion.
* Patients with hypo- or hyperthyroidism as determined by history, or screening TSH results.
* Patients with known or suspected perforation or obstruction.
* History of gastric retention, inflammatory bowel disease, bowel resection, or colostomy.
* Patients with a known history of organic cause for their constipation.
* Patients meeting the ROME definition of Irritable Bowel Syndrome
* Patients currently taking any of the following medications that are known to effect bowel habits:

  * Antidiarrheals
  * Antacids containing magnesium or aluminum salts
  * Anticholinergics
  * Antispasmodic agents
  * Erythromycin and other macrolides
  * Octreotide
  * Lotronex, Zofran, or other 5-HT3 antagonists
  * Zelnorm, or other 5-HT4 agonists
  * Opiods/narcotic analgesics
  * Prokinetics
  * Serotonin re-uptake inhibitors or tricyclic antidepressants
  * Calcium antagonists
* Patients who are breastfeeding, pregnant, or intend to become pregnant during the study.
* Female patients of childbearing potential who refuse a pregnancy test.
* Patients with a known allergy to polyethyleneglycol.
* Patients who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Patients who, within the past 30 days have participated in an investigational clinical study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-07; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse events and laboratory testing)

SECONDARY OUTCOMES:
Assessment of constipation using ROME I criteria and analysis of individual ROME I criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Herrera, MD, Principal Investigator — University of South Alabama
Locations (43):
- United States (43):
  - Hoover, Alabama
  - Mobile, Alabama
  - Pell City, Alabama
  - Tallassee, Alabama
  - Glendale, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Sacramento, California
  - Washington D.C., District of Columbia
  - Kissimmee, Florida
  - Lake Worth, Florida
  - Largo, Florida
  - Ocoee, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Oakbrook Terrace, Illinois
  - Peoria, Illinois
  - Overland Park, Kansas
  - Laurel, Maryland
  - Springfield, Massachusetts
  - St Louis, Missouri
  - South Bound Brook, New Jersey
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Greer, South Carolina
  - Bristol, Tennessee
  - Kingsport, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - Salt Lake City, Utah
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia